CLINICAL TRIAL: NCT01294852
Title: A Randomized Trial: Comparison of Two Strategies for Surfactant Prophylaxis in Premature Infants
Brief Title: Comparison of Two Strategies for Surfactant Prophylaxis in Premature Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Ankara University Faculty of Medicine, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ankara University-01; Ankara University (Other Grant/Funding Number: Ankara University Research Fund (Number 10B3330010))
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2009-12

CONDITIONS: Premature Birth; Premature Lungs
Keywords: prophylactic; surfactant; premature; mechanical ventilation; mortality; morbidities
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate bolus surfactant (Experimental)
  Interventions: Other: surfactant prophylaxis
- post-resuscitation surfactant (Experimental)
  Interventions: Other: surfactant prophylaxis

INTERVENTIONS:
Other: surfactant prophylaxis — Premature infants born before 28 weeks' gestation and infants born at 29 to 30 weeks' gestation who did not receive antenatal steroid were randomized before delivery to receive either immediate bolus or post-resuscitation surfactant prophylaxis at 15 minutes after birth. Those infants who were randomized to immediate bolus surfactant were intubated as rapidly as possible after birth, were administered 100 mg/kg surfactant (Curosurf[Chiesi, Farmaceutici, Parma, Italy]), and received standard resuscitation measures as indicated. Those infants who were randomized to post-resuscitation surfactant received standard resuscitation measures first, were intubated electively at 15 minutes after birth and received 100 mg/kg surfactant (Curosurf[Chiesi, Farmaceutici, Parma, Italy]).

SUMMARY:
The purpose of this study is to determine whether the immediate bolus strategy combined with early nasal CPAP (nCPAP) treatment could decrease the subsequent need for ventilation compared to the administration of surfactant prophylaxis at 15 minutes after birth with early nCPAP in premature infants.

DETAILED DESCRIPTION:
Respiratory distress syndrome (RDS) is a syndrome in premature infants caused by developmental insufficiency of surfactant production and structural immaturity in the lungs. Exogenous surfactant therapy has become well established in newborn infants with RDS. Surfactant replacement therapy, either as a rescue treatment or a prophylactic, reduces mortality and several aspects of morbidity in babies with RDS. It is known that infants who are at a significant risk of RDS should receive prophylactic surfactant therapy, but the optimal timing and strategy for prophylactic surfactant therapy remains controversial. When administered immediately after delivery, surfactant mixes with the fetal lung fluid and reaches the alveoli before the onset of lung injury potentially created by the first applied positive pressure ventilation. As another approach, surfactant prophylaxis may be administered after resuscitation and stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born before 28 weeks' gestation
* Premature infants born at 29 to 30 weeks' gestation who did not receive antenatal steroid were randomized before delivery

Exclusion Criteria:

* Infants died at delivery room

Ages: 1 Minute to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
ventilatory requirement | within the first 5 days of life
  Infants with RDS may require mechanical ventilation. Mechinal ventilation causes volu- and barotrauma in the lungs and associated morbidities. The earlier surfactant is given, the better it works. So immediate surfactant prophylaxis given before the first breath may decrease the requirement for mechanical ventilation compared with surfactant prophylaxis given at 15 minutes of age after resuscitation and stabilization.

SECONDARY OUTCOMES:
Pneumothorax | first 72 hours of life
Pulmonary hemorrhage | first 72 hours of life
patent ductus arteriosus | first one week
necrotizing enterocolitis | first one month
retinopathy of prematurity | first two months
intraventricular hemorrhage | first one week
bronchopulmonary dysplasia | first two months
duration of hospitalization | one year
mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Arsan, Professor, Study Director — Ankara University Faculty of Medicine; Emel Okulu, MD, Principal Investigator — Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine Department of Pediatrics, Ankara, Turkey (Türkiye)